CLINICAL TRIAL: NCT03082183
Title: Effects of Rifampicin on the Pharmacokinetics of BI 425809 Following Oral Administration in Healthy Male Subjects (an Open-label, Two-period, Fixed-sequence Trial)
Brief Title: A Study in Healthy Men to Test Whether Rifampicin Influences the Amount of BI 425809 in the Blood
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1346-0018; 2016-004862-24 (EudraCT Number)
Record Dates: First submitted 2017-03-10; First posted 2017-03-17 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Healthy
MeSH Terms: interventions — Rifampin; BI 425809

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All participants (Experimental): BI 425809 given alone in first period, then in combination with Rifampicin in second period
  Interventions: Drug: Rifampicin; Drug: BI 425809

INTERVENTIONS:
Drug: Rifampicin — once daily
Drug: BI 425809 — once daily
  Other Names: Iclepertin

SUMMARY:
The primary objective of this trial is to investigate the relative bioavailability of a single dose of BI 425809 when given alone (Reference, B) compared with co-administration (Test, A) on the 7th day of a 10-day treatment with rifampicin following oral administration in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, based on a complete medical history including a physical examination, vital signs (Blood Pressure (BP), Pulse Rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 55 years (incl.)
* BMI of 18.5 to 29.9 kg/m2 (incl.)
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and local legislation

Exclusion Criteria:

* Any finding in the medical examination (including Blood Pressure (BP), Pulse Rate (PR) or Electrocardiogram (ECG)) is deviating from normal and judged as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy and/or surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy and simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Use of drugs within 30 days prior to administration of trial medication if that might reasonably influence the results of the trial (incl. QT/QTc interval prolongation)
* Participation in another trial where an investigational drug has been administered within 60 days prior to planned administration of trial medication, or current participation in another trial involving administration of investigational drug
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking on specified trial days
* Alcohol abuse (consumption of more than 20 g per day)
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days prior to administration of trial medication or intended donation during the trial
* Intention to perform excessive physical activities within one week prior to administration of trial medication or during the trial
* Inability to comply with dietary regimen of trial site
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because considered not able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study

In addition, the following trial-specific exclusion criteria apply:

* History of relevant liver diseases such as disturbance of liver function, jaundice, drug induced liver injury, Dubin-Johnson syndrome, Rotor syndrome, or liver tumours
* Thrombocytes below lower limit of normal or liver enzymes (Alanine transaminase (ALT), Aspartate transaminase (AST), Gamma-Glutamyl trsanspeptidase (GGT), Alkaline phosphatase (AP)) above upper limit of normal at the screening examination

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2017-03-28 (Actual); Primary Completion 2017-06-20 (Actual); Study Completion 2017-06-20 (Actual)

PRIMARY OUTCOMES:
AUC0-168 (area under the concentration-time curve of BI 425809 in plasma over the time interval from 0 to 168 h) | up to 168 hours
  AUC0-168 (area under the concentration-time curve of BI 425809 in plasma over the time interval from 0 to 168 h)
Cmax (maximum measured concentration of BI 425809 in plasma) | up to 51 days
  Cmax (maximum measured concentration of BI 425809 in plasma)

SECONDARY OUTCOMES:
AUC0-∞ (area under the concentration-time curve of BI 425809 in plasma over the time interval from 0 extrapolated to infinity) | up to 51 days
  AUC0-∞ (area under the concentration-time curve of BI 425809 in plasma over the time interval from 0 extrapolated to infinity)
t1/2 (terminal half-life of BI 761036 in plasma) | up to 51 days
  t1/2 (terminal half-life of BI 761036 in plasma)

CONTACTS AND LOCATIONS:
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany

REFERENCES:
- [Derived] Desch M, Wunderlich G, Goettel M, Goetz S, Liesenfeld KH, Chan TS, Rosenbrock H, Sennewald R, Link J, Keller S, Wind S. Effects of Cytochrome P450 3A4 Induction and Inhibition on the Pharmacokinetics of BI 425809, a Novel Glycine Transporter 1 Inhibitor. Eur J Drug Metab Pharmacokinet. 2022 Jan;47(1):91-103. doi: 10.1007/s13318-021-00723-y. Epub 2021 Oct 29. PMID 34716565

DOCUMENTS (2):
  • Study Protocol (2017-04-05): https://cdn.clinicaltrials.gov/large-docs/83/NCT03082183/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-21): https://cdn.clinicaltrials.gov/large-docs/83/NCT03082183/SAP_001.pdf